CLINICAL TRIAL: NCT05897996
Title: Percutaneous Anastomosis Creation for Hemodialysis Access
Acronym: PACHA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties with the device
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-PP-22; 2022-A01847-36 (Other: ANSM)
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: D001159
Keywords: vascular access for hemodialysis; Arterio-Arterial Fistula
MeSH Terms: conditions — Arterio-Arterial Fistula | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- creation of vascular access for hemodialysis (Experimental): creation of vascular access for hemodialysis with percutaneous AVF creation
  Interventions: Device: creation of vascular access for hemodialysis

INTERVENTIONS:
Device: creation of vascular access for hemodialysis — endo-AVfs created with Wavelinq

SUMMARY:
The investigators propose to adult patients needing the creation of a vascular access for hemodialysis, not eligible to the creation of a distal AVF, to create a percutaneous anastomosis between an artery and a vein (endo-AVFs). The study is a prospective single-center cohort (Nice University Hospital) with a 2-year follow-up (recruitment: 18 months, length of study per patient: 24 months, data analysis: 6 months). After the procedure, patients will receive duplex-ultrasound follow-up, according to local practice, at 6 weeks (+ surgical examination), 3, 6, 12, 18 and 24 months.

DETAILED DESCRIPTION:
1. Inclusion baseline Visit The patient is adressed by his/her nephrologist for the creation of a vascular access for hemodialysis. It is provided with a venous and arterial map of the two upper limbs (not specific to the study) as well as a blood test necessary for anesthesia.
2. Inclusion visit The patient is examined by the vascular surgeon who determines, via arterial and venous mapping, and once the inclusion and non-inclusion criteria have been reviewed, whether he is eligible for the study. Participation in the protocol is then proposed to him. If he agrees to participate, the patient signs the informed consent after an appropriate time for reflection.

   The anesthesia consultation and the date of the procedure are scheduled during this visit.
3. Response: V0 The patient is hospitalized in the vascular surgery department, preferably in the day surgery unit, or in the full hospitalization department if he lives too far away or cannot be accompanied.

   Once in the operating room, and after anesthetic induction, the surgeon proceeds to create the percutaneous fistula. At the end of the intervention, the surgeon performs the shivering and the patient goes back to the service or remains for a while in the post-operative monitoring room depending on the anesthesia he has received.

   The patient is allowed to go home the same day for UCA patients, or the next day for patients on full hospitalization; once the surgeon has verified the presence of the thrill and the absence of signs of early ischemia, characterized or hematomas.

   The patient leaves with his appointment date at 6 weeks.
4. Follow-up to S6: V1

   The patient is seen again 6 weeks after the operation. The consultation begins with a Doppler to determine:
   * Permeability of access
   * The absence of venous and arterial stenosis
   * The flow in the humeral artery
   * The internal diameter of the vein and artery 2cm from the anastomosis
   * Good distal hand perfusion

   The patient then sees the surgeon who proceeds:
   * The presence of thrill
   * The absence / presence of hematomas, lymphocele
   * Signs of venous hypertension
   * Signs of neurological deficit
   * Vascular steal syndrome This consultation (Doppler and surgical follow-up) is done routinely for all creations of fistulas and is not specific to the study.

   If the vascular access is ready to be used, the surgeon indicates the possible puncture points on the map obtained from the Doppler. The date of first dialysis is noted by the nephrologist.

   During the first 5 sessions, the nephrologist informs:

   The type of needle
   * Who performs the puncture
   * The use of ultrasonographic guidance to perform the puncture

   The nephrologist completes a satisfaction questionnaire at the end of the first dialysis session (as well as at 3, 6, 12, 18 and 24 months after the access was created). This questionnaire includes 5 items: ease of vein palpation, ease of vein puncture, appearance of the arm with respect to their prior experience, quality of dialysis and their overall satisfaction.
5. Monitoring at M3, M6, M12, M18 and M24: visits V2 to V6 The following visits contain a Doppler (identical to that carried out in V1 and included in the routine management of the patient) the results of which may lead to a consultation with the surgeon depending on the results.

It is recommended that vascular access flow be measured monthly. The months without Doppler, it will be measured during dialysis sessions (according to Transonic or Dialysance depending on the equipment of the dialysis center).

The frequency of the Dopplers will be adjusted if necessary in the event of reoperation and the opinion of the surgeon may be requested.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient referred by the nephrologist for the creation of a vascular access for hemodialysis
* Patient eligible for the creation of an arteriovenous fistula of the upper limb further to assessment by the surgeon
* Pre-operative venous and arterial Doppler ultrasound performed on the upper limbs, the results of which meet the following criteria for the same limb:

  * Perforating vein present and permeable, with no stenosis, measuring at least 2 mm in diameter
  * Permeable cephalic vein of the arm, rectilinear over at least 10 cm, with no stenosis, measuring at least 2.5 mm
  * Permeable ulnar and/or radial vein, with no stenosis, measuring at least 2 mm in diameter
  * Permeable ulnar and/or radial vein, with no stenosis or major calcifications, measuring at least 2 mm in diameter
  * Permeable brachial artery, with no stenosis, with no major calcifications
* Informed consent signature (by the designated trusted person if necessary)
* Membership of a social security system

Exclusion Criteria:

* History of vascular access for hemodialysis on the same limb (except for a distal radiocephalic fistula with chronic malfunction or dialysis catheter)
* Patients eligible for the creation of a distal vascular access, at the anatomical snuffbox or the wrist, with the following criteria:

  1. Clinical examination of the upper limbs highlighting a cephalic vein at the distal 1/3 of the forearm, a radial pulse, an ulnar pulse and a negative Allen test, and
  2. Pre-operative venous and arterial Doppler ultrasound performed on the upper limbs, showing:

     * a permeable cephalic vein on the forearm, with no stenosis, measuring at least 2 mm in diameter at the distal 1/3 of the forearm over a length of at least 15 cm.
     * a permeable radial artery, with no stenosis, with no major calcifications, measuring at least 2 mm in diameter at the distal 1/3 of the forearm, not dominant,
     * a permeable ulnar artery, with no stenosis nor calcifications,
     * a permeable palmar arch, functional, with no stenosis or calcifications
* Patients treated with immunosuppressants
* Patients having had or scheduled to have major surgery in the six weeks prior or further to inclusion
* Patients with radial arterial and/or ulnar artery thrombosis
* Patients with a vascular anomaly, including a target artery-vein distance that is too great or a venous or arterial thrombosis that is pre-existing or discovered on the day of the procedure, which does not permit use of the device.
* Patients with a severe known allergy to iodinated contrast agents
* Patients under guardianship or trusteeship
* Patients deprived of freedom
* Pregnant patients (women of child-bearing age will receive a urine pregnancy test to rule out pregnancy prior to inclusion, results will be given to them by the doctor of their choosing).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
to assess the maturation rate of endo-Arterio venous fistula created with Wavelinq | at 3 months
  assessed as the ratio between the number of successful maturation of the access at 3 month and the total number of Arterio venous fistula created

SECONDARY OUTCOMES:
nephrologist's satisfaction. | 3 months.
  complete a satisfaction questionnaire
nephrologist's satisfaction. | 6 months.
  complete a satisfaction questionnaire
nephrologist's satisfaction. | 12 months.
  complete a satisfaction questionnaire
nephrologist's satisfaction. | 18 months.
  complete a satisfaction questionnaire
nephrologist's satisfaction. | 24 months.
  complete a satisfaction questionnaire
To assess the primary patency of Arterio venous fistula created percutaneously | 1 year
  defined by the length of time in months between Arterio venous fistula creation and 1) any later surgery or procedures aiming to rectify or restore Arterio venous fistula function OR 2) abandonment of the Arterio venous fistula
To assess the primary patency of Arterio venous fistula created percutaneously | 2 years
  defined by the length of time in months between Arterio venous fistula creation and 1) any later surgery or procedures aiming to rectify or restore AVF function OR 2) abandonment of the Arterio venous fistula

CONTACTS AND LOCATIONS:
Overall Officials: Nirvana SADAGHIANLOO, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, CHU de NICE, France

IPD SHARING:
Plan to Share IPD: No